CLINICAL TRIAL: NCT01794390
Title: Critical Errors in Pulmojet and Other Devices
Brief Title: Handling Inhalers - Technique Error Comparison (HI-TEC)
Acronym: HI-TEC
Status: Completed | Type: Observational
Sponsor: Research in Real-Life Ltd (Network)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, David Price, Prof., MD, Professor of Primary Care Respiratory Medicine (University of Aberdeen) and Managing Director of Research in Real-Life Ltd., Research in Real-Life Ltd
Other Study IDs: PJ1201
Record Dates: First submitted 2013-02-14; First posted 2013-02-18 (Estimated); Last update posted 2015-10-27 (Estimated); Status verified 2015-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Asthma
Keywords: COPD (Chronic Obstructive Pulmonary Disease); Asthma; Pulmojet; Inhalers; Respiratory; Inhaler Technique; Critical Errors
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Turbuhaler and MDI patients (Arm 1): Patients (Diskus naive) will be randomised to receive training on the PulmoJet© device followed by Diskus, or vice versa
- Diskus patients (Arm 2): Patients (Turbuhaler naive) will be randomised to receive training on the PulmoJet© device followed by Turbohaler, or vice versa

SUMMARY:
Randomised, cross sectional, observational study evaluating inhaler device critical errors (errors that could affect dose delivery to the lungs) for the Pulmojet inhaler compared to Diskus or Turbuhaler in asthma and COPD patients receiving regular maintenance inhaled steroid therapy.

DETAILED DESCRIPTION:
Single-visit, randomised, crossover, open-label study comparing critical device handling errors for the Pulmojet compared to Diskus with Turbohaler in patients receiving maintenance inhaled corticosteroid (ICS) or ICS plus long acting beta2 agonist via Diskus, Turbuhaler or pMDI. Pulmojet is an inhaler developed by Zentiva (a subsidiary of Sanofi Aventis); other inhalers are the major prescribed inhalers in the treatment of asthma and COPD. This will allow critical errors in the use of the Pulmojet inhaler to be assessed and evaluated against commonly prescribed inhalers.

376 patients recruited from 10 primary care practices will be invited to participate in this single visit study. Upon entry to the study, all patients will be assessed as to their current inhaler device technique before entering into a randomised cross-over to receive device training according to their current device:

Current Diskus users (i.e. Turbuhaler naive): will be randomised to receive inhaler device training for the Pulmojet device followed by the Turbuhaler, or vice versa.

Current Turbuhaler / pMDI users (i.e. Diskus naive): will be randomised to receive inhaler device training for the Pulmojet device followed by the Diskus, or vice versa.

For all devices, critical errors in the use of inhalers will be assessed through nurse observation and vitalograph pneumotrac spirometry ('technology recorded'). A two step device training protocol will be used to establish the ease to which patients can be taught to use the study devices (Pulmojet, Turbohaler (in current Diskus users) and Diskus (in current Turbohaler or pMDI users). In Step 1 patients will be given the product Patient Information Leaflet (PIL) to read, and in Step 2 patients will be asked to watch a device instructional video. After each step patients will be assessed on their device use. Patients will progress from Step 1 to Step 2 unless device mastery is achieved at Step 1, in which case the patient will progress onto the second device or the study will have been completed.

All inhalers provided to participants will be supplied completely empty, i.e. with no active drug or placebo present, and participants will not receive any medication or interventional procedure during the study conduct.

An independent virtual steering committee has been assembled to oversee the study protocol. The steering committee members are international inhalation technology experts.

The primary objective will be to evaluate the critical errors and number of steps to achieve device mastery (defined as absence of critical errors):

* Diskus vs. Pulmojet
* Turbuhaler vs. Pulmojet

The secondary objective will be to evaluate critical errors in device use between:

• Current device vs. Pulmojet (all patients)

ELIGIBILITY:
Inclusion Criteria:

1. Patient is aged over 18
2. Patient has an asthma and/ or COPD diagnosis
3. Patient is receiving current therapy including either inhaled corticosteroids (ICS) or fixed dose combination ICS/ Long acting Beta-agonists(FDC ICS/LABA's)
4. The patient's current therapy is being administered through a metered dose inhaler (MDI), Turbuhaler or Diskus device
5. Patients must be able and willing to read and comprehend written and verbal instructions
6. After full explanation, patients must have signed an informed consent document indicating that they understand the purpose of and the procedures required for the study and are willing to participate in the study
7. All Turbuhaler and MDI patients are required to have no use of the Diskus device in the past year
8. All Diskus patients are required to have no use of the Turbuhaler device in the past year

Exclusion Criteria:

1. Current therapy with ICS or ICS/LABA in any device other than a Diskus, Turbuhaler or metered dose inhaler (MDI)
2. An acute or chronic condition that, in the investigator's opinion, would limit the patient's ability to participate in this study
3. Patient has received oral steroids and/or antibiotics for a lower respiratory condition (identified using lower respiratory diagnoses) in the 4 weeks preceding the study (used as a proxy measure for identifying an exacerbation and / or lower respiratory infection, which might suggest altered inspiratory capabilities)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from a representative UK primary care asthma and COPD population
Sampling Method: Probability Sample
Enrollment: 431 (Actual)
Dates: Start 2013-09; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Nurse-observed critical inhaler technique errors | up to 1 year
  Proportion of patients making errors considering nurse-observed errors only with Pulmojet vs comparator. Comparator was Diskus for current Turbuhaler and MDI patients, and Turbuhaler for current Diskus patients.
  A maximum of 2 attempts is allowed (self taught using a patient information leaflet (PIL), patient video).
  A list of critical errors for each inhaler has been produced by an independent steering committee.
  Nurse observed critical errors are recorded using a device-specific error checklist.

SECONDARY OUTCOMES:
All critical inhaler technique errors (including both nurse-observed and inhalation errors recorded via the Vitalograph Pneumotrac Spirometer) | up to 1 year
  All critical inhaler technique errors (including both nurse-observed and inhalation errors recorded via the Vitalograph Pneumotrac Spirometer). Proportion of patients making errors considering all critical inhaler technique errors was compared between 1) Pulmojet vs comparator and 2) Pulmojet vs current device. Comparator was Diskus for current Turbuhaler and MDI patients, and Turbuhaler for current Diskus patients.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. David Price, Investigator, Study Director — Research in Real Life
Locations (1):
- UK GP sites, Cambridge, United Kingdom

REFERENCES:
- [Background] Gupta R, Sheikh A, Strachan DP, Anderson HR. Burden of allergic disease in the UK: secondary analyses of national databases. Clin Exp Allergy. 2004 Apr;34(4):520-6. doi: 10.1111/j.1365-2222.2004.1935.x. PMID 15080802
- [Background] Molimard M, Le Gros V. Impact of patient-related factors on asthma control. J Asthma. 2008 Mar;45(2):109-13. doi: 10.1080/02770900701815727. PMID 18350401
- [Background] Haughney J, Price D, Barnes NC, Virchow JC, Roche N, Chrystyn H. Choosing inhaler devices for people with asthma: current knowledge and outstanding research needs. Respir Med. 2010 Sep;104(9):1237-45. doi: 10.1016/j.rmed.2010.04.012. Epub 2010 May 15. PMID 20472415
- [Background] Price D, Thomas M. Breaking new ground: challenging existing asthma guidelines. BMC Pulm Med. 2006 Nov 30;6 Suppl 1(Suppl 1):S6. doi: 10.1186/1471-2466-6-S1-S6. PMID 17140424
- [Background] Thomas M, Price D. Impact of comorbidities on asthma. Expert Rev Clin Immunol. 2008 Nov;4(6):731-42. doi: 10.1586/1744666X.4.6.731. PMID 20477123
- [Background] Giraud V, Roche N. Misuse of corticosteroid metered-dose inhaler is associated with decreased asthma stability. Eur Respir J. 2002 Feb;19(2):246-51. doi: 10.1183/09031936.02.00218402. PMID 11866004
- [Background] Molimard M, Raherison C, Lignot S, Depont F, Abouelfath A, Moore N. Assessment of handling of inhaler devices in real life: an observational study in 3811 patients in primary care. J Aerosol Med. 2003 Fall;16(3):249-54. doi: 10.1089/089426803769017613. PMID 14572322
- [Background] Haughney J, Price D, Kaplan A, Chrystyn H, Horne R, May N, Moffat M, Versnel J, Shanahan ER, Hillyer EV, Tunsater A, Bjermer L. Achieving asthma control in practice: understanding the reasons for poor control. Respir Med. 2008 Dec;102(12):1681-93. doi: 10.1016/j.rmed.2008.08.003. Epub 2008 Sep 23. PMID 18815019
- [Derived] Chrystyn H, Price DB, Molimard M, Haughney J, Bosnic-Anticevich S, Lavorini F, Efthimiou J, Shan D, Sims E, Burden A, Hutton C, Roche N. Comparison of serious inhaler technique errors made by device-naive patients using three different dry powder inhalers: a randomised, crossover, open-label study. BMC Pulm Med. 2016 Jan 14;16:12. doi: 10.1186/s12890-016-0169-5. PMID 26769482
- See also: Organisation's webpage — http://www.optimumpatientcare.org/
- See also: U.K. Webpage providing information on Asthma — http://www.asthma.org.uk/
- See also: Organisation's webpage — http://www.rirl.org